CLINICAL TRIAL: NCT03209596
Title: Nutritional and Biochemical Effects of Orange Juice Supplementation in Soccer Players: a Double Blind, Randomized and Controlled Trial
Brief Title: Orange Juice Supplementation in Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ellen Cristini de Freitas (Other)
Collaborators: Citrosuco Company (Industry)
Responsible Party: Sponsor-Investigator, Ellen Cristini de Freitas, PhD, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ECdeFreitas
Record Dates: First submitted 2017-06-21; First posted 2017-07-06 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Healthy Athletes
Keywords: Athletes; Food intake; Supplementation; Biochemical biomarkers; Soccer Players

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All assignments and group randomization were performed by a research team member who was not directly involved in the study. The masking of the volunteers was performed by the control drink. For statistical analysis of the results, the masking was maintained by conferring fictitious names to the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orange juice (Experimental): Seventeen individuals received 1 liter/day of pasteurized orange juice. Participants consumed the orange juice before and post exercise, the volume of juice per serving was 500 mL. On players' rest days, the juice was consumed throughout the day.
  Interventions: Dietary Supplement: Orange juice (1L/d)
- Control drink (Active Comparator): Thirteen individuals received 1 liter/day of control drink. The participants consumed the control drink before and post exercise, the volume of drink per serving was 500 mL. On players' rest days, the drink was consumed throughout the day. The control drink consisted of an aqueous solution containing sucrose (44 g), glucose (22 g), fructose (22 g), citric acid (11g) (proportionally 2:1:1:0.5) (USDA, 2016) (with the same proportion of total sugars as the orange juice, and without all others bioactive compounds of juice), dyestuff sunset yellow (0.05 g) and orange essence.
  Interventions: Dietary Supplement: Control drink (1L/d)

INTERVENTIONS:
Dietary Supplement: Orange juice (1L/d) — The players (n=17) drank 1 liter per day of orange juice. We do not interfere on the volunteers' usual diet during the study, and they did not ingest any commercial nutritional supplements in this period. During the intervention, the volunteers were engaged in a common training routine specified by the coach's team.
  Arms: Orange juice
Dietary Supplement: Control drink (1L/d) — The players (n=13) drank 1 liter per day of the control drink during a 60-day period. We do not interfere on the volunteers' usual diet during the study, and they did not ingest any commercial nutritional supplements in this period. During the intervention, the volunteers were engaged in a common training routine specified by the coach's team.
  Arms: Control drink

SUMMARY:
This study aimed to verify if orange juice supplementation can be a nutritional strategy to ensure an adequate energy and micronutrients ingestion, influencing metabolic responses of soccer players.

DETAILED DESCRIPTION:
Thirty-four male soccer players aged 18.5 ± 0.5 years and BMI (Body Mass Index) of 21.41 ± 1.48 kg/cm2 were randomly divided into two parallel groups: (1) orange juice (n = 17), composed of individuals receiving 1 liter/day of orange juice; (2) control (n = 17) composed of individuals receiving 1 liter/day of control drink with the same proportion of total sugars as the orange juice. The recruitment process began in September 2013, the intervention was carried out from November 2013 to January 2014, and the data analysis started in February 2014. The sample size took into account the variances in total cholesterol, considering the high statistical variability of biochemical markers, which requires a sufficient number of samples to ensure representativeness and adequate statistical power of analysis, and that the reduction of total cholesterol is associated to the regular consumption of orange juice (Dourado et al., 2015). Based on unpublished data from a previous pilot experiment, it was expected that the total cholesterol of orange juice group would be 10% lower in relation to control group after intervention (orange juice = 123.41 ± 12.12 mg/dL, control drink = 37.80 ± 11.17 mg/dL). Thus, with a type I error α = 0.05 and a type II error β = 0.2 (80% power) the minimum sample size should have 12 individuals per group (n = 24). Considering the high layoffs rate in the team, the initial sample size of study was constituted by 17 individuals per group (n = 34). During the intervention, four individuals from control drink group failed the study protocol, and the study was concluded with 30 participants (orange juice n = 17 and control drink n = 13). Primary and secondary endpoints were the improvement of food intake and changes in biochemical markers, respectively. Shapiro Wilk and Levene tests evaluated normality and homogeneity of data, respectively. T-test was conducted to identify possible differences between groups at baseline. A mixed factorial ANOVA was applied to determine the effect of treatment and time, within and between groups (Sidak post hoc test), and statistical significance was set at p < 0.05. Food intake, biochemical biomarkers and body composition were assessed before and after the 60 days of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Three consecutive years of soccer training prior to the start of the study.

Exclusion Criteria:

* Historic of chronic disease, use of hormones, drugs, vitamins supplements and/or other dietary supplements during the study.

Ages: 18 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2013-10-20 (Actual); Primary Completion 2014-01-31 (Actual); Study Completion 2014-08-29 (Actual)

PRIMARY OUTCOMES:
Food intake | 60 days
  Food intake was assessed by 24-hour recall

SECONDARY OUTCOMES:
Glucose | 60 days
  Blood dosing using commercial kits
Glycated hemoglobin | 60 days
  Blood dosing using commercial kits
Total cholesterol | 60 days
  Blood dosing using commercial kits
Low Density Lipoprotein Cholesterol (LDL-C) | 60 days
  Calculated with an equation described by Friedewald et al. (1972)
High Density Lipoprotein Cholesterol (HDL-C) | 60 days
  Blood dosing using commercial kits
Triglycerides | 60 days
  Blood dosing using commercial kits
Creatinine | 60 days
  Blood dosing using commercial kits

OTHER OUTCOMES:
Body Mass Index (BMI kg/cm2) | 60 days
  Weight and height will be combined to report BMI (kg/cm2) by the following equation: BMI (kg/cm2) = Weight (kg) / (Height (m))2
% Lean body mass | 60 days
  Assessed by deuterium oxide method
% Fat body mass | 60 days
  Assessed by deuterium oxide method
% body water | 60 days
  Assessed by deuterium oxide method

CONTACTS AND LOCATIONS:
Overall Officials: Ellen C De Freitas, Ph.D., Principal Investigator — University of São Paulo, School of Physical Education and Sports of Ribeirão Preto; Sara M Terrazas, Msc, Study Chair — Sao Paulo State University "Julio de Mesquita Filho", Faculty of Pharmaceutical Sciences
Locations (1):
- University of São Paulo, School of Physical Education and Sports of Ribeirão Preto., Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedewald WT, Levy RI, Fredrickson DS. Estimation of the concentration of low-density lipoprotein cholesterol in plasma, without use of the preparative ultracentrifuge. Clin Chem. 1972 Jun;18(6):499-502. No abstract available. PMID 4337382
- [Result] Dourado GK, Cesar TB. Investigation of cytokines, oxidative stress, metabolic, and inflammatory biomarkers after orange juice consumption by normal and overweight subjects. Food Nutr Res. 2015 Oct 20;59:28147. doi: 10.3402/fnr.v59.28147. eCollection 2015. PMID 26490535